CLINICAL TRIAL: NCT02831309
Title: Active Class Space Metabolic Benefits Study
Acronym: ACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Rebecca Hasson, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00084540
Record Dates: First submitted 2016-06-29; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Childhood Obesity
Keywords: physical activity
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sedentary Condition (Sham Comparator): Forty minutes of screen time. Standardized meals provided.
  Interventions: Behavioral: Sedentary Condition
- Light-Intensity Condition (Active Comparator): Forty minutes of light-intensity activity. Standardized meals provided.
  Interventions: Behavioral: Light-Intensity Condition
- Moderate-Intensity Condition (Active Comparator): Forty minutes of moderate-intensity activity. Standardized meals provided.
  Interventions: Behavioral: Moderate-Intensity Condition
- High-Intensity Condition (Active Comparator): Forty minutes of high-intensity activity. Standardized meals provided.
  Interventions: Behavioral: High-Intensity Condition

INTERVENTIONS:
Behavioral: Light-Intensity Condition — The light-intensity condition consisted of 8 hours of sitting interrupted with 2--minute, light--intensity activity breaks performed at 25% of heart rate reserve (HRR) every 18 minutes. Standardized meals were provided.
  Arms: Light-Intensity Condition
Behavioral: Moderate-Intensity Condition — The moderate-intensity condition consisted of 8 hours of sitting interrupted with 2--minute, moderate-intensity activity breaks performed at 50% of heart rate reserve (HRR) every 18 minutes. Standardized meals were provided.
  Arms: Moderate-Intensity Condition
Behavioral: High-Intensity Condition — The high-intensity condition consisted of 8 hours of sitting interrupted with 2--minute, vigorous-intensity activity breaks performed at 75% of heart rate reserve (HRR) every 18 minutes. Standardized meals were provided.
  Arms: High-Intensity Condition
Behavioral: Sedentary Condition — The sedentary condition consisted of 8 hours of sitting interrupted with 2-minutes of screen time every 18 minutes. Standardized meals were provided.
  Arms: Sedentary Condition

SUMMARY:
ACS examined the potential influence of intermittent physical activity breaks of various intensities (control, light, moderate, vigorous) on measures of immediate mental performance, mood, hunger and several metabolic outcomes in children aged 7-11 years. We build upon previous work to hypothesize that higher-intensity intermittent physical activity breaks throughout an 8-hour day will improve immediate mental performance, mood, and post-exercise physical activity levels, while reducing hunger and post-exercise food intake.

DETAILED DESCRIPTION:
Background: A range of metabolic, behavioral, mental and physical health benefits of regular physical activity have been documented in adults and children in the long-term. Yet, relatively little is known about how children's usual daily physical activity patterns (i.e. small bursts throughout the day) affect acute (immediately post-activity) and short-term (72 hours post-activity) metabolic and psychosocial outcomes. Additionally, little is known how this specific pattern of physical activity affects subsequent physical activity levels (i.e. compensatory behavior) and subsequent dietary intake, over the short-term- information critical to designing effective interventions involving the physical environment of the school classroom. Overall Goal: Active Class Space (ACS) will examine the potential influence of intermittent physical activity breaks of various intensities (control, light, moderate, vigorous) on measures of immediate mental performance, mood, hunger and several metabolic outcomes in children aged 7-11 years. We build upon previous work to hypothesize that higher-intensity intermittent physical activity breaks throughout an 8-hour day will improve immediate mental performance, mood, and post-exercise physical activity levels, while reducing hunger and post-exercise food intake. Specific Aims: (1) To determine the effects of intermittent physical activity breaks of varying intensities on immediate mental performance, hunger and satiety; (2) To determine the effects of intermittent activity breaks of varying intensities on ratings of perceived exertion (RPE), perceived exercise enjoyment, in-task mood, post-exercise food intake and post-exercise physical activity levels; and (3) To examine gender differences in the preceding variables in response to low-, moderate, and high-intensity intermittent physical activity. Design: Eighteen healthy males and twenty-one healthy females between the ages of 7-11 years completed completed four experimental conditions in random order: (1) 8 hours of sitting interrupted with 2--minute, light--intensity activity breaks performed at 25% of heart rate reserve (HRR) every 18 minutes; (2) 8 hours of sitting interrupted with 2--minute, moderate--intensity activity breaks (50% HRR); (3) 8 hours of sitting interrupted with 2--minute, high--intensity activity breaks (75% HRR); and (4) 8 hours of sitting interrupted with 2 minutes of sedentary screen time. Standardized meals will be provided during each experimental condition. Dietary intake and physical activity levels were monitored for the remainder of the experimental day and over the subsequent three days for each condition. Dependent Variables: Major outcome variables include: Energy expenditure measured by indirect calorimetry and heart rate; dietary intake measured using a 3-day dietary record; physical activity measured by accelerometry; immediate mental performance assessed using a 90-sec mathematical computation test; hunger and satiety assessed using a visual analog scale; RPE assessed using the Borg scale; perceived exercise enjoyment assessed using the physical activity enjoyment scale (PACES); in-task mood assessed using the Feeling Scale (FS) and Subjective Exercise Experiences Scale (SEES). Data Analysis: A linear mixed model will be fitted for each outcome variable with effects for condition, sex, BMI, and baseline physical activity level. A Bonferroni correction will be used to adjust for multiple comparisons in post hoc tests following the mixed-effect model. A similar linear mixed-model for raw levels of each outcome variable over time will also be fitted to assess temporal differences between conditions. This model will include effects for condition, time, time-by-condition interaction, sex, BMI, and baseline physical activity levels. Significance: ACS will shed new light on the short-term metabolic, behavioral, mental and physical health benefits of intermittent physical activity breaks in children. The results from this study will inform the design of behavioral and environmental interventions to promote physical activity and cognitive development in pediatric populations.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 7-11 years old from the greater Ann Arbor and Ypsilanti areas were recruited to participate in this study.

Exclusion Criteria:

* Participants were excluded based on the following criteria: (1) were taking medications or were diagnosed with diseases that could influence exercise ability or cognitive function and (2) were previously diagnosed with any major illness/health condition since birth.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Physical activity energy expenditure | 4 days
  Physical activity energy expenditure throughout the condition day and over the next three days. Participants wore an accelerometer for four days. Energy expenditure was calculated from accelerometer data.

SECONDARY OUTCOMES:
40-item immediate mental performance math test | 1 day
  Number of math questions answered correctly within 90 seconds in the morning (800hr), midday (1200hr) and afternoon (1600hr). Scores were marked as number correct out of 40.
Dietary intake | 4 days
  Standardized meals were provided in the morning, midday and evening and 3-day dietary records were collected three days post-condition day. Total daily dietary intake was calculated from food consumed in the lab and at home.
Physical activity minutes | 4 days
  Physical activity minutes throughout the condition day and over the next three days. Participants wore an accelerometer for four days. Minutes participating in physical activity was calculated using accelerometer data.
4-item hunger and satiety visual analog scale | 1 day
  Self reported hunger and satiety in the morning (800hr), midday (1200hr) and afternoon (1600hr). Scores were calculated from a visual analog scale ranging from 0-100 (0= hungry; 0=full), yielding a total between 0- 400
Single-item ratings of perceived exertion | 1 day
  Perceived exertion during 20, 2-minute activity or sedentary breaks. This single item questionnaire is scored 6-20 (6 = light exertion; 20 maximal exertion).
Single-item feeling scale | 1 day
  Participants self-reported how they felt during each 20, 2-minute activity or sedentary breaks. This single item questionnaire is scored -5 to +5 (-5 = very bad; +5 = very good).
16-item exercise enjoyment measure | 1 day
  Self-reported mood in the morning (800hr), midday (1200hr) and afternoon (1600hr). The scale is a combination of 16 positive and negative statements. The responses were scored on a 5-point Likert like scale (1= disagree a lot, 5 = agree a lot). Seven of the 16 statements were reverse scored.
12-item psychological mood measure | 1 day
  Self-reported mood at midday (1200hr) and afternoon (1600hr). A 3 dimensional, 12-item scale designed to measure changes in 3 categories; positive well-being (e.g., i feel terrific), psychological distress (e.g., i feel miserable), and fatigue (e.g., i feel exhausted). For each item participants will be asked to indicate how strongly they are experiencing the feeling state at that time. Items will be scored on a 7-point Likert scale (1 = "not at all," 7 = "very much so"). Each subscale ranges from 4 to 28 with higher scores representing greater fatigue, positive well-being or psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca E Hasson, PhD, Principal Investigator — University of Michigan
Locations (1):
- Childhood Disparities Research Laboratory, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weston E, Nagy M, Ajibewa TA, O'Sullivan M, Block S, Hasson RE. Acute Effects of Interrupting Prolonged Sitting With Intermittent Physical Activity on Blood Pressure in Preadolescent Children. Pediatr Exerc Sci. 2019 Nov 1;31(4):408-415. doi: 10.1123/pes.2018-0224. Epub 2019 Jun 27. PMID 30849931
- [Derived] Block SS, Tooley TR, Nagy MR, O'Sullivan MP, Robinson LE, Colabianchi N, Hasson RE. Acute Effect of Intermittent Exercise and Action-Based Video Game Breaks on Math Performance in Preadolescent Children. Pediatr Exerc Sci. 2018 Aug 1;30(3):326-334. doi: 10.1123/pes.2017-0183. Epub 2018 Feb 27. PMID 29485933
- [Derived] Nagy MR, O'Sullivan MP, Block SS, Tooley TR, Robinson LE, Colabianchi N, Hasson RE. Affective Responses to Intermittent Physical Activity in Healthy Weight and Overweight/Obese Elementary School-Age Children. J Phys Act Health. 2017 Nov 1;14(11):845-851. doi: 10.1123/jpah.2016-0552. Epub 2017 Oct 6. PMID 28682697
- [Derived] O'Sullivan MP, Nagy MR, Block SS, Tooley TR, Robinson LE, Colabianchi N, Hasson RE. Acute Compensatory Responses to Interrupting Prolonged Sitting With Intermittent Activity in Preadolescent Children. Pediatr Exerc Sci. 2018 May 1;30(2):259-265. doi: 10.1123/pes.2017-0078. Epub 2017 Oct 12. PMID 28605263